CLINICAL TRIAL: NCT05208125
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Safety, Tolerability and Immunogenicity Study of Candidate HIV-1 Vaccines ChAdOx1.HTI and MVA.HTI With Recombinant HIV-1 Envelope Protein ConM SOSIP.v7 gp140 Vaccine, Adjuvanted With MPLA Liposomes in ART-Suppressed HIV-1 Positive Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IrsiCaixa (Other)
Collaborators: José Moltó Marhuenda, PhD, MD (Unknown); Beatriz Mothe Pujadas PhD,MD (Unknown); Susana Benet Garrabé, PhD,MD (Unknown); Lucía Bailón Álvarez, MD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCN03
Record Dates: First submitted 2021-11-03; First posted 2022-01-26 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HIV Infection
Keywords: Human immunodeficiency; Virus; Vaccine; HIV; Safety; Tolerability
MeSH Terms: conditions — HIV Infections; Virus Diseases | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either the combined regimen with T- and B-cell immunogens (CSSMS) or placebo (PPPPP) in a double-blinded fashion at a ratio of 2:1.
Who Masked: Participant, Investigator
Masking Description: Upon preparation, masking of the study products will take place in the same preparation room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSSMS (Experimental): ChAdOx1.HTI at week 0, ConM SOSIP.v7 at weeks 4, 12 and 28, and MVA.HTI at week 22 (CSSMS).
  Interventions: Biological: ChAdOx1.HTI at week 0, ConM SOSIP.v7 at weeks 4, 12 and 28, and MVA.HTI at week 22 (CSSMS).
- PPPPP (Placebo Comparator): Normal saline solution at weeks 0, 4, 12, 22, and 28 (PPPPP).
  Interventions: Other: Normal saline solution

INTERVENTIONS:
Biological: ChAdOx1.HTI at week 0, ConM SOSIP.v7 at weeks 4, 12 and 28, and MVA.HTI at week 22 (CSSMS). — Intramuscular administration of 1 x ChAdOx1.HTI (5x1010 Vp), 3 x ConM SOSIP.v7 (100μg) adjuvanted with MPLA liposomes (500μg), and 1 x MVA.HTI (2x108pfu)
  Arms: CSSMS
Other: Normal saline solution — Intramuscular administration of normal saline solution
  Arms: PPPPP

SUMMARY:
BCN03 is a Single-site, randomized, double-blind, placebo-controlled, phase I study to evaluate the safety, tolerability, immunogenicity, and efficacy of a vaccine regimen that includes a sequence of the T- and B-cell immunogens ChAdOx1.HTI and MVA.HTI and ConM SOSIP.v7 gp140 adjuvanted with MPLA liposomes in 30 virologically-suppressed ART-treated HIV-1 positive individuals.

DETAILED DESCRIPTION:
Participants will be randomized to receive either the combined regimen with T- and B-cell immunogens (CSSMS) or placebo (PPPPP) in a double-blinded fashion at a ratio of 2:1. Safety and immunogenicity of the combined T- and B-cell regimen will be measured up to week 30 (2 weeks after last ConM SOSIP.v7/placebo administration). At week 30, all participants will undergo an ATI of 24 weeks of duration. At visit week 54 (End-of-ATI visit), or before according to pre-specified criteria, ART will be resumed. Efficacy endpoints will be measured at 12 and 24 weeks of ATI (study visits week 42 and 54). After ART resumption, participants will be followed during an additional safety period of 12 weeks (study visit week 66, End-of-Study visit). Treatment allocation will remain blinded until week 54 (End-of-ATI visit).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged at least 18 years on the day of screening and no greater than 60 years on the day of the first IMP administration.
2. Confirmed HIV-1 infection.
3. Optimal virological suppression for at least 2 years prior to the screening visit, defined as maintained pVL <50 cop/ml allowing for isolated blips (non-consecutive 50-200 copies/mL)
4. Being on the same ART regimen within at least 4 weeks prior to screening visit.
5. CD4 count ≥ 500 cells/mm3 at the screening visit.
6. Nadir CD4 count ≥ 350 cells/mm3. Lower counts at the moment of acute HIV-1 infection will be allowed only if appropriate immune recovery was followed after ART initiation and ART was not initiated within first 6 months after estimated time of HIV-1 acquisition.
7. Willing and able to be adherent to their ART regimen for the duration of the study.
8. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
9. In the opinion of the Principal Investigator or designee, the candidate has understood the information provided and capable of giving written Informed Consent.
10. If heterosexually active female of childbearing potential(1), using an effective method of contraception (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner(1) from 14 days prior to the first IMP administration and commit to use it until four months after the last IMP administration or until her pVL is <50 copies/mL in two-consecutive determinations after ART resumption, whichever is later. All female candidates of childbearing potential who are not heterosexually active at screening, must agree to utilise an effective method of contraception if they become heterosexually active during the study.
11. If heterosexually active male, regardless of reproductive potential, sterilized or agree on the use of an effective method of contraception by his female partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility(2) from the day of the first IMP administration until four months after the last IMP administration or until his pVL is <50 copies/mL in two-consecutive determinations after ART resumption, whichever is later. All male candidates who are not heterosexually active at screening, must agree to utilise an effective method of contraception if they become heterosexually active during the study.
12. Il female, willing to undergo urine pregnancy tests at the designated time points.
13. Willing to accept blood draws and collect stool at time points specified in the Schedule of Events (Appendix VII).
14. Willing to forgo donating blood, eggs, or sperm from the first IMP administration until four months after last IMP administration or until his or her pVL is <50 copies/mL in two-consecutive determinations after ART resumption, whichever is later.

    * (1) A woman will be considered of childbearing potential if not permanently sterilized nor postmenopausal. Permanent sterilization methods include tubal ligation, hysterectomy and bilateral oophorectomy. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
    * (2) Condom use nor diaphragm are considered as an additional method of contraception only and cannot be the only method of contraception used as not been considered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Exclusion Criteria:

1. If female, pregnant or planning a pregnancy during the study and until at least four months after the last IMP administration or until her pVL is <50 copies/mL in two-consecutive determinations after ART resumption, whichever is later; or lactating.
2. ART initiated within 6 months from the estimated time of HIV-1 acquisition documented by immediate ART initation after a) an HIV-1 documented seroconversion (<180 days), b) an HIV-1 diagnose with negative or indeterminate western blot test or positive p24 antigenemia and/or c) presenting with symptoms suggestive of acute retroviral syndrome.
3. When available, pre-ART genotypic data that demonstrates the presence of clinically significant drug resistance mutations that could prevent the construction of a viable ART regimen post-treatment interruption.
4. Reported periods of suboptimal adherence to ART or suboptimal ART regimens (dual therapy allowed as switch-regimens if sustained viral uppression pVL<50 copies/ml is documented).
5. History of past ART interruptions longer than 2 weeks.
6. Participation in another clinical trial that involves a treatment intervention (active arm) within 12 weeks of study entry (at screening visit).
7. Any AIDS-defining disease or progression of HIV-related disease.
8. History of autoimmune disease.
9. History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study.
10. Receipt of approved vaccines within 3 weeks of study entry(1)
11. Known hypersensitivity to any component of the IMP formulation, or severe or multiple allergies to drugs or pharmaceutical agents.
12. Previous immunisation with any experimental immunogens.
13. Potential participant received or plans to receive:

    1. licensed live attenuated vaccines - within 28 days before or after planned administration of the first or subsequent study vaccinations. For details regarding COVID-19 vaccines, see bullet c and d below.
    2. other licensed (not live) vaccines - within 14 days before or after planned administration of the first or subsequent study vaccinations. For details regarding COVID-19 vaccines, see bullet c and d below.
    3. Recombinant viral vectored COVID-19 vaccines or live attenuated COVID-19 vaccines, either licensed or authorized for emergency use (eg. Emergency Use Authorization [EUA], Emergency Use Listing [EUL] or similar program) - within 28 days before or after planned administration of the first or subsequent study vaccinations.
    4. Other COVID-19 vaccines than the ones specified in bullet c (eg. mRNA vaccines, protein-based vaccines) either licensed or authorized for emergency use (eg. EUA, EUL or similar program) - within 14 days before or after planned administration of the first or subsequent study vaccinations.
14. Receipt of blood products within 3 months of study entry.
15. Treatment for cancer or lymphoproliferative disease within 1 year of study entry.
16. Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents (use on inhaled steroids for asthma or topic steroids for localized skin conditions are permitted).
17. Any other current or prior therapy which, in the opinion of the investigator, would make the individual unsuitable for the study or influence the results of the study.
18. Any laboratory abnormalities including:

    Hematology
    * Hemoglobin < 10.0 g/dl
    * Absolute Neutrophil Count ≤ 1,000 /mm3 (≤ 1 x 109/L)
    * Absolute Lymphocyte Count ≤ 600 /mm3 (≤ 0.6 x 109/L)
    * Platelets ≤100,000 /mm3, ≥ 550,000 /mm3 (≤ 100 /L, ≥ 550 /L) Biochemistry
    * Creatinine > 1.3 x ULN
    * Aspartate aminotransferase (AST) > 2.5 x ULN
    * Alanine aminotransferase (ALT) > 2.5 x ULN

    Microbiology
    * Positive for hepatitis B surface antigen,
    * Positive for hepatitis C antibody, unless confirmed clearance of HCV infection (spontaneous or following treatment)
    * Positive serology indicating active syphilis requiring treatment(2)
19. Refusal to an eventual ART interruption within the scope of the study objectives(3).

    * (1)Efforts will be made to ensure all participants included are updated on their Hepatitis A, Hepatitis B and Pneumococcal vaccinations before enrolment. Seasonal Flu vaccinations or other required vaccinations will be scheduled to avoid the 3 weeks preceding and following IMP administrations and the first 12 weeks of ATI.
    * (2) Cases in which positive RPR titres are detected but syphilis has been confirmed to have been properly treated will be allowed into the study if treatment has been given >4 weeks prior to study entry/IMP administration.
    * (3)A questionnaire related to ART interruption will be answered by the candidate during the screening visit to be able to address Expectations and Worries in a timely manner to reduce the risk of participants lost to follow-up during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Local IMP-related AEs of Grade 3 and 4 | From first administration up to week 30 (i.e., start of ATI, 2 weeks after last administration).
  Proportion of participants that develop Grade 3 or 4 local IMP-related AEs, based on the DAIDS scale
Systemic IMP-related AEs of Grade 3 and 4 | From first administration up to week 30 (i.e., start of ATI, 2 weeks after last administration).
  Proportion of participants that develop Grade 3 or 4 systemic IMP-related AEs, based on the DAIDS scale
Descriptive of AEs | From first administration up to week 30 (i.e., start of ATI, 2 weeks after last administration)
  Descriptive summary of any local and systemic AEs, including laboratory abnormalities, severity, durability, and relationship to IMP in vaccine recipients.

SECONDARY OUTCOMES:
De novo T-cell Immunogenicity to HTI | From week 0 to week 30
  Proportion of participants who develop de-novo T-cell responses to HTI- during the intervention period as determined by IFN (gamma) ELISPOT.
Magnitude, focus and breadth of T-cell Immunogenicity to HTI | From week 0 to week 30
  Magnitude, focus and breadth of HTI-specific T-cell responses during the intervention period as determined by IFN (gamma) ELISPOT
B-cell Immunogenicity (serum titers of NAbs) | From week 0 to week 30
  Serum titers of autologous neutralizing antibodies (NAbs) during the intervention period
B-cell Immunogenicity (proportion of NAbs) | From week 0 to week 30
  Proportion of participants with autologous NAbs during the intervention period
B-cell Immunogenicity (magnitude of trimer binding antibodies) | From week 0 to week 30
  Magnitude of trimer binding antibodies during the intervention period
B-cell Immunogenicity (proportion of trimer binding antibodies) | From week 0 to week 30
  Proportion of participants with a trimer binding antibody response during the intervention period
B-cell Immunogenicity (serum titers heterologous neutralising antibodies) | From week 0 to week 30
  Serum titres of heterologous neutralising antibodies (i.e., against additional [Tier 1a/b, Tier 2] virus strains) during the intervention period
B-cell Immunogenicity (proportion of heterologous neutralising antibodies) | From week 0 to week 30
  Proportion of participants with heterologous neutralising antibodies during the intervention period
Viral rebound during ATI (sustained viral remission) | At 12 and 24 weeks after ATI start
  Percentage of participants with sustained viral remission, defined as pVL <50 copies/mL at 12 and 24 weeks after ATI start, respectively
Viral rebound during ATI (time to viral detection) | From ATI start to the first occurrence of detectable pVL pVL (from week 30 to week 54 (ATI period)
  Time to viral detection, defined as the time from ATI start to the first occurrence of detectable pVL (≥50 copies/mL).
Viral rebound during ATI (post-rebound viral control) | At 12 and 24 weeks after ATI start
  Percentage of participants with post-rebound viral control, defined as a pVL <2,000 copies/mL at 12 and 24 weeks after ATI start, respectively
Viral rebound during ATI (percentage of off-ART) | At 12 and 24 weeks after ATI start
  Percentage of participants who remain off-ART at 12 and 24 weeks after ATI start, respectively.
Viral rebound during ATI (time off-ART) | From ATI start to ART resumption (from week 30 to week 54 (ATI period)
  Time off-ART, defined as time from ATI start to ART resumption.
Safety of an ATI period (symptoms compatible with acute retroviral syndrome) | From week 30 to week 54
  Proportion of participants who develop symptoms compatible with acute retroviral syndrome
Safety of an ATI period (stress/anxiety related to ATI) | From week 30 to week 54
  Proportion of participants with clinically significant changes in the ATI Psychological questionnaire suggestive of stress/anxiety related to ATI.
Safety of an ATI period (seeking of psychological support) | From week 30 to week 54
  Proportion of participants who seek psychological support during and/or after ATI.
Safety of post-ATI ART resumption (viral suppression) | From week 54 to week 66
  Proportion of participants who suppress pVL to <50 copies/mL 12 weeks after ART resumption.
Safety of post-ATI ART resumption (new mutations conferring clinically-significant resistance to antiretroviral drugs) | From week 54 to week 66
  Proportion of participants who develop new mutations not present in the pre-ART viral genotype conferring clinically-significant resistance to antiretroviral drugs. In those participants not reaching viral re-suppression 12 weeks after ART resumption, an ART viral genotype will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain